CLINICAL TRIAL: NCT06964568
Title: Concurrent Chemoradiotherapy Followed by PD-1 Inhibitor Maintenance Therapy in Locally Advanced Esophageal Squamous Cell Carcinoma: a Randomized Phase III Trial
Brief Title: CCRT Followed by PD-1 Inhibitor Maintenance Therapy in Locally Advanced ESCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai 27
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Carcinoma; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Immune Checkpoint Inhibitors; Radiotherapy; TP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCRT and PD-1 inhibitor maintenance therapy (Experimental): Radiotherapy: 50.4Gy/28Fx. Chemotherapy: Paclitaxel 135mg/m2 d1+cisplatin 25mg/m2 d1-3 q28d
  PD-1 inhibitors will be administered intravenously, a fixed dose of 200 mg, once every 3 weeks for 1 year within 42 days after the end of radiotherapy
  Interventions: Drug: PD-1 inhibitor; Radiation: Radiotherapy; Drug: TP regimen
- CCRT and surveillance (Active Comparator): Radiotherapy: 50.4Gy/28Fx. Chemotherapy: Paclitaxel 135mg/m2 d1+cisplatin 25mg/m2 d1-3 q28d
  Interventions: Radiation: Radiotherapy; Drug: TP regimen

INTERVENTIONS:
Drug: PD-1 inhibitor — PD-1 inhibitors will be administered intravenously, a fixed dose of 200 mg, once every 3 weeks for 1 year.
  Arms: CCRT and PD-1 inhibitor maintenance therapy
Radiation: Radiotherapy — Radiotherapy 50.4Gy/28Fx
Drug: TP regimen — Chemotherapy: Paclitaxel 135mg/m2 d1+cisplatin 25mg/m2 d1-3 q28d

SUMMARY:
The goal of this clinical trial is to learn if concurrent chemoradiotherapy followed by immunotherapy as maintenance therapy works to treat locally advanced esophageal squamous cell cancer in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged 18 years or above
3. Histologically confirmed esophageal squamous cell carcinoma
4. Clinical stages T3-4N0M0 or TxN+M0 or TxNxM1 (Only for supraclavicular lymph nodes) based on the 8th UICC-TNM classification

7. Eastern Cooperative Oncology Group(ECOG) performance status: 0-1 8. Life expectancy ≥3 months 9. Adequate organ functions Absolute neutrophil counts (ANC) ≥1.5×109⁄L; Hemoglobin (Hb) ≥9g⁄dl; Platelet (Plt) ≥100×109⁄L; Total bilirubin ≤1.5 upper limit of normal (ULN); Aspartate transaminase (AST) ≤2.5 ULN; Alanine aminotransferase (ALT) ≤2.5 ULN; Creatinine ≤1.5 ULN

Exclusion Criteria:

1. Esophageal perforation or hematemesis
2. Any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism and hypothyroidism (effective hormone replacement therapy excepted)) and immunosuppressive agents or systemic hormonal therapy indicated within 28 days (for adverse events of chemoradiotherapy excepted).
3. Previously received or receiving PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1.
4. Allergic to any of the ingredients in PD-1 inhibitors for injection.
5. Uncontrolled heart diseases or clinical symptoms, such as: (1) New York Heart Association(NYHA) class II or higher heart failure; (2) unstable angina; (3) myocardial infarction within 1 year; (4)clinically significant arrhythmia requiring clinical intervention.
6. Congenital or acquired immunodeficiency (such as HIV infection); active hepatitis B (HBV-DNA≥104 copy number/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method); active tuberculosis.
7. Active infection or unexplained fever >38.5 °C within 2 weeks before randomization (fever due to tumor excepted, according to investigator).

   Patients with fertility reluctant to take contraceptive measures during the trial, or female patients pregnant or breastfeeding.
8. According to the investigator, other factors that may cause termination of the study. ie, other serious diseases (including mental illness) require combined treatment, family or social factors, which may affect the safety or the collection of trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  PFS for all patients with PD-1 inhibitor maintenance therapy vs all patients with surveillance

SECONDARY OUTCOMES:
PFS | 2 years
  PFS for TDLN-sparing RT followed by PD-1 inhibitor maintenance therapy vs TDLN-sparing RT followed by surveillance
OS | 2 years
Adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided